CLINICAL TRIAL: NCT03120780
Title: High Dose Epidural Fentanyl for Second Stage Labor Analgesia
Brief Title: Epidural Fentanyl for 2nd Stage Labor Analgesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to change on standard of care, higher doses of fentanyl requirements are rare.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Goran Ristev, Assistant Professor - Clinical, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016H0439
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl; Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two groups: one group will receive lower dose epidural fentanyl (20 micrograms) combined with local anesthetic; and one group will receive higher-dose epidural fentanyl (100micrograms) combined with the same amount of local anesthetic.
Who Masked: Participant
Masking Description: The subject and the research personnel will be blinded to the arm to which they are randomized. Only the clinician assessing the patient and administering epidural doses will be not be blinded to the study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Dose Fentanyl (Active Comparator): Low dose epidural fentanyl combined with local anesthetic as 10mL of 0.125% bupivacaine with 20 mcg fentanyl (Fentanyl 20 mcg)
  Interventions: Drug: Fentanyl 20 mcg
- High Dose Fentanyl (Experimental): High dose epidural fentanyl combined with local anesthetic as 10mL of 0.125% bupivacaine with 100 mcg fentanyl (Fentanyl 100 mcg)
  Interventions: Drug: Fentanyl 100 mcg

INTERVENTIONS:
Drug: Fentanyl 20 mcg — 20 mcg fentanyl in 10 mL 0.125% bupivacaine
  Other Names: Low Dose
  Arms: Low Dose Fentanyl
Drug: Fentanyl 100 mcg — 100 mcg fentanyl in 10 mL 0.125% bupivacaine
  Other Names: High Dose
  Arms: High Dose Fentanyl

SUMMARY:
This study is being done to investigate if there is more effective pain relief during the latter stages of labor and delivery when epidural fentanyl 100mcg is administered compared to epidural fentanyl 20mcg.

DETAILED DESCRIPTION:
The objective is to evaluate if high-dose epidural fentanyl (100 micrograms) is more effective at providing pain relief during the late first stage (>8 cm cervical dilation) and second stage of labor until the time of delivery compared to low-dose epidural fentanyl (20 micrograms). In this study, anesthetic care will be provided to a subject by an experienced anesthesia provider according to standard hospital care. If the subject has adequate pain relief from the continuous epidural infusion, then a study investigator will record the verbal pain score and document any other side effects at hourly intervals beginning at >8cm cervical dilation, but no additional epidural medications will be administered. If pain relief becomes inadequate during the late first or second stage of labor (>8cm cervical dilation) and a manual epidural bolus is required, then the subject will be randomly assigned to one of two groups (like flipping a coin): one group will receive lower dose epidural fentanyl (20 micrograms) combined with local anesthetic; and one group will receive higher-dose epidural fentanyl (100micrograms) combined with the same amount of local anesthetic. Both doses are used frequently on labor and delivery and are considered to be safe based on available evidence. If there is not sufficient pain relief from the epidural medication given, then an experienced anesthesia provider will assess if another epidural dose may be effective and this additional epidural medication will be given at the discretion of the anesthesia provider. An experienced anesthesia provider will be available at all times during the study to assess pain and provide epidural medications. All patients participating in the study will have their pain scores assessed every hour as soon as the cervical dilation is noted to be >8cm; at the time of randomization; and at 10, 20, 30 and 60 minutes after the epidural dose is administered. The presence of any side-effects such as itching, shivering, nausea, vomiting, low blood pressure, slow respiratory rate or lower extremity muscle weakness will also be collected at hourly intervals as soon as the cervical dilation is noted to be >8cm. Subject satisfaction (1-100 rating scale) with anesthetic care provided will be assessed on postpartum day # 1 during routine follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women
2. Spontaneous labor
3. A single vertex presentation fetus at term (38-42 weeks)
4. Effective labor epidural analgesia with continuous epidural infusion established
5. Provide written consent to participate in the study.

Exclusion Criteria:

1. Multigravida women
2. Multigestation pregnancies
3. Patients being treated/managed for chronic pain
4. Allergies or significant adverse reactions to local anesthetic or opioid medications
5. Inadequate or unsatisfactory labor epidural analgesia
6. Patients with history of spine abnormalities or spine surgery
7. Non-English speaking
8. Prisoners
9. Age less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be pregnant woman to considered for study.
Enrollment: 65 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
VRS Pain Score | 30 minutes after epidural bolus
  VRS Pain score

SECONDARY OUTCOMES:
VRS Pain Score | At Time of Delivery
  VRS Pain Score
Mode of Delivery | At Time of Delivery
  Mode of Delivery (cesarean, spontaneous vaginal or assisted vaginal delivery)
Patient Satisfaction | During labor until post-partum day one
  Patient Satisfaction with Labor Pain Control (1-100 rating scale; 1= not satisfied at all, 100=completely satisfied)
Adverse Events | During labor until post-partum day one
  Nausea, vomiting, shivering, pruritis, hypotension, motor block, maternal respiratory depression, neonatal outcomes
Rescue Epidural Boluses | Until delivery
  Total number of clinician administered epidural boluses during the late first (≥8cm cervical dilation) and second stages of labor

CONTACTS AND LOCATIONS:
Overall Officials: John Coffman, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.